CLINICAL TRIAL: NCT03695445
Title: A Prospective Study of the Safety of Norepinephrine Administered Through Peripheral Venous Catheter During Surgery
Brief Title: Safety of Norepinephrine Administered Through Peripheral Venous Catheter
Status: Completed | Type: Observational
Sponsor: Christer Svensen (Other)
Responsible Party: Sponsor-Investigator, Christer Svensen, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: EudraCT2018-002158-59; 2018-002158-59 (EudraCT Number)
Record Dates: First submitted 2018-09-14; First posted 2018-10-04 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Peripheral Norepinephrine: Patients who will undergo surgery with need for vasopressor support.
  Interventions: Drug: Peripheral administration of Norepinephrine

INTERVENTIONS:
Drug: Peripheral administration of Norepinephrine — Systematic follow-up of complications from peripheral administration of Norepinephrine

SUMMARY:
Norepinephrine is a drug that elevates the blood pressure. It is routinely administered through peripheral catheters during surgery. There is a risk of tissue damage in case of leakage of Norepinephrine from the catheter to the surrounding tissue. Another risk is irregular administration of Norepinephrine due to kinking of the peripheral catheter. This could lead to fluctuations in blood pressure. The primary aim of the study is to investigate complications from Norepinephrine administered in peripheral venous catheters. The secondary aim is to investigate if comorbidity, placement of the peripheral catheter or the duration of the infusion are associated with a higher rate of complications. 1000 patients will be included. Inclusion criteria: Patients who will undergo surgery with need for vasopressor support. Exclusion criteria: The patient has a central venous catheter, a peripherally inserted central venous catheter or lack of informed consent.

DETAILED DESCRIPTION:
In many hospitals in Sweden, Norepinephrine is administered through peripheral venous catheters in the operating room. However there are very few studies to support the safety of peripherally administered Norepinephrine.

Norepinephrine of the concentration 8 respectively 40 microg/ml will be investigated. The primary aim of the study is to investigate complications from Norepinephrine administered in peripheral venous catheters. The secondary aim is to investigate if comorbidity, placement of the peripheral catheter or the duration of the infusion are associated with a higher rate of complications.

The localisation and size of the peripheral venous catheter will be registered. The blood pressure will me measured every 5 minutes and every minute in case of systolic blood pressure over 220 mm Hg.

The site of administration will regularly be monitored for complications. If subcutaneous infusion of Norepinephrine is suspected, the patient will be followed up for up to 48 hours or until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has general anesthesia or central blocks
* Need for vasopressors in the pre, per or postoperative period to maintain adequate mean arterial blood pressure
* Age ≥18 years

Exclusion Criteria:

* The patient has a central venous line
* The patient has a peripherally inserted central line
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who require vasopressors to maintain an adequate blood pressure during general anesthesia and/or central blocks.
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with treatment-related adverse events | 0-72 hours
  Proportion of patients with complications (Subcutaneous infusion and/or hypertension>220 mmHg and/or heart rate<40 beats/min)

SECONDARY OUTCOMES:
Association between comorbidity, placement of catheter, duration of infusion and increased proportion of complications | 0-72 hours
  Odds ratio of Treatment-Emergent Adverse Events in risk groups (ASA>2, placement of catheter distal to the antecubital or popliteal fossae, duration of infusion> 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Andersson, MD, Principal Investigator — Stockholm South General Hospital
Locations (3):
- Sweden (3):
  - Danderyds sjukhus, Stockholm, Danderyd
  - Södersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No